CLINICAL TRIAL: NCT06103331
Title: Surveillance for Invasive Fungal Infections in Selected Hospitals in Dhaka City, Bangladesh
Brief Title: Fungal Surveillance in Bangladesh
Status: Recruiting | Type: Observational
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Institute of Epidemiology, Disease Control and Research (Other)
Responsible Party: Sponsor
Other Study IDs: PR-21142
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Invasive Fungal Infections
Keywords: Invasive Fungal Pathogen; Hospitalized patients; Surveillance
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- child: identification and management of invasive fungal pathogen
  Interventions: Other: Invasive Fungal disease surveillance
- adult: identification and management of invasive fungal pathogen
  Interventions: Other: Invasive Fungal disease surveillance

INTERVENTIONS:
Other: Invasive Fungal disease surveillance — Management of invasive fungal infection according to pathogen identification and susceptibility report.

SUMMARY:
This will be an exploratory descriptive study designed to conduct surveillance for the identification of invasive fungal pathogens among hospitalized patients in Bangladesh at two tertiary care acute-level hospitals. including the Dhaka Medical College Hospital, the Dhaka Hospital of icddr,b, and the National Institute of Cancer Research Hospital (NICRH). Respiratory samples, blood, urine, cerebrospinal fluid, surgical wound infection swabs, and other samples including biopsy tissue specimens will be obtained at intensive care units, general medicine and surgery wards, post-operative care, etc. The collected specimens will be sent to the clinical microbiology laboratories of the surveillance hospitals or to the pathology laboratory (biopsy tissue specimens) to test for Aspergillus, Histoplasms, Candida, Pneumocystis, Cryptococcus, and Mucormycetes. The lab. methods will include microscopy, staining, culture, and biochemical tests mainly and if feasible then some specimens may undergo molecular or immunological methods.

DETAILED DESCRIPTION:
1. Burden:

   Over 300 million people worldwide are infected with a deadly fungal infection, with 25 million at high risk of death or blindness. Population and disease demographics are used to calculate the worldwide burden of fungal diseases (age, gender, HIV infection, asthma, etc).

   Given the growing number of immunocompromised individuals especially among hospitalized patients who are at increased risk for invasive fungal infections, fungal illnesses require more attention than ever before. The importance of fungal diseases contributing to worldwide morbidity and mortality is emphasized. To assess the burden of these diseases more precisely, long-term, sustainable monitoring systems for fungal diseases, as well as better noninvasive and reliable diagnostic methods, are required.

   Even though most deaths from fungal illnesses are preventable, they are still a neglected topic by public health authorities. Other health issues, such as asthma, AIDS, cancer, organ transplantation, and corticosteroid therapy, can result in serious fungal infections. Antifungal therapy can be started right away if a correct diagnosis is made early. Recent global estimates have found 3,000,000 cases of chronic pulmonary aspergillosis, ~223,100 cases of cryptococcal meningitis complicating HIV/AIDS, ~700,000 cases of invasive candidiasis, ~500,000 cases of Pneumocystis jirovecii pneumonia, ~250,000 cases of invasive aspergillosis, ~100,000 cases of disseminated histoplasmosis, over 10,000,000 cases of fungal asthma and ~1,000,000 cases of fungal keratitis occur annually.
2. Knowledge gap:

Currently, there is no ongoing national surveillance system to detect invasive fungal pathogens or serious health threats. Hence, there is inadequate data on the burden, types, and diversity of fungal species in particular among hospitalized patients in Bangladesh. Some noteworthy issues affecting the proper diagnosis of invasive fungal pathogens in Bangladesh are an inadequate number of trained laboratory personnel to diagnose fungal diseases, only a few healthcare facilities performing fungal culture, insufficient awareness about severe fungal infections, lack of prioritization for fungal disease surveillance in healthcare delivery, lack of understanding about utilization of surveillance data to guide diagnosis and treatment, lack of antifungal drug stewardship and diagnostic stewardship and significant logistical challenges to ensure adequate biosecurity for diagnosis of and prevention against severe fungal infections.

Relevance:

Investigators need to take the necessary steps that will gradually lead to the establishment of a national surveillance system for invasive fungal pathogens, increase the generation of country-representative fungal surveillance data, improve surveillance data usage and reporting, and enhance IPC activities in Bangladesh.

Objectives:

To identify hospitalized patients infected with invasive fungal pathogens.

Description of the research project:

Methods:

This will be an exploratory descriptive study designed to conduct surveillance for the identification of invasive fungal pathogens among hospitalized patients in Bangladesh at two tertiary care acute-level hospitals.

The primary outcomes to be measured in this study:

The proportion of laboratory-identified invasive fungal pathogens among hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

Must include all of the following criteria:

1. Admitted/hospitalized patients of any age and gender in tertiary-level acute care hospitals AND
2. Having any of the following co-morbid immunosuppressive conditions or risk factors for healthcare-associated fungal infections such as:

   * Chronic lung conditions including asthma, COPD
   * Hemodialysis patients,
   * diabetes,
   * Patients receiving chemotherapy or immunosuppressive drugs (e.g. corticosteroids, immunosuppressive drugs among organ transplant recipients), for ≥7 days
   * Patients with AIDS
   * Patients at risk of healthcare-associated infections (e.g., Patients under postoperative care, having a urinary catheter, with tracheal intubation, under ventilatory support, secured with intravenous (IV) cannula, any other invasive procedures, etc.)
   * Hospitalized Patients under prolonged injectable antibiotic treatment (>7 days)
   * Prolonged hospitalization more than 7 days.
   * History of taking steroids or antibiotics for more than 2 weeks prior to hospitalization

   AND
3. Patients or caregivers providing consent

For children aged <5 years, the age criteria and additional inclusion criteria will be as follows:

* 0 to 59-month-old children of either sex admitted in hospital with any illness.
* Have features of sepsis/pneumonia (based on clinical features below)

And any of the following criteria:

* Those who will fail to respond to injectable antibiotics or both 1st and 2nd line antibiotics (1st line- inj. Ampicillin plus gentamicin, 2nd line- inj. Ceftriaxone plus levofloxacin/gentamicin as per icddr,b hospital protocol)
* Any child with SAM or h/o recent measles or any condition that may induce immune suppression plus fail to respond to injectable antibiotics/ 1st line antibiotics (1st line antibiotics- inj. Ampicillin +inj. Gentamicin)
* Those who will develop late-onset hospital-associated infection (LOHAI)
* Any child who will require ICU care for more than 7 days
* Develop extensive thrush after taking long-term injectable antibiotics
* History of taking steroids or antibiotics for more than 2 weeks prior to hospitalization

Exclusion Criteria:

* History of taking antifungal drugs within 2 weeks
* Not willing to give consent

Min Age: 0 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients meeting the inclusion criteria and having ONE of the following groups of clinical features suggestive of infection of a particular organ system during sample collection:
  * Clinical features suggestive of infection of the respiratory system:
    * Fever or chills WITH
    * Cough or shortness of breath WITH
    * Abnormal lung findings on chest auscultation or on chest X-ray or CT scans
  * Clinical features of sepsis:
    * Hyperthermia or hypothermia (rectal temperature >38.5 Celsius or <35 Celsius respectively) and tachycardia plus either bounding pulses or, altered mental status or, hypoxemia in absence of pneumonia or, abnormal WBC count (>12×109 ⁄ L or, <4 ×109 ⁄ L or, band and neutrophil ratio ≥ 0.1) or, increased serum lactate level (diagnosed by physicians)
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of laboratory-identified invasive fungal pathogens among hospitalized patients. | July 2022 - September 2026
  The primary goal will be to ensure a sustainable surveillance platform in low-income settings such as Bangladesh. The Investigators will utilize four strategies to establish a sustainable fungal surveillance platform/program in Bangladesh which will be as follows:
  1. Increase capacity to conduct surveillance
  2. Identify and respond
  3. Target and train
  4. Monitor, evaluate and improve

CONTACTS AND LOCATIONS:
Overall Officials: Sayeeda Huq, MBBS,MIPH, Principal Investigator — International Centre for Diarrheal Diseases Research, Bangladesh
Locations (1):
- International Centre for Diarrheal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No